CLINICAL TRIAL: NCT04982081
Title: Treating Congestive Heart Failure Patients With Human iPSC-derived Cardiomyocytes Through Catheter-based Endocardial Injection
Brief Title: Treating Congestive HF With hiPSC-CMs Through Endocardial Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Help Therapeutics (Industry)
Collaborators: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTao
Record Dates: First submitted 2021-07-01; First posted 2021-07-29 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases; Congestive Heart Failure; Dilated Cardiomyopathy
Keywords: induced pluripotent stem cell; Congestive heart failure; Regenerative medicine; dilated cardiomyopathy
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hiPSC-CM therapy low dosage (Experimental)
  Interventions: Biological: hiPSC-CM therapy
- hiPSC-CM therapy high dosage (Experimental)
  Interventions: Biological: hiPSC-CM therapy

INTERVENTIONS:
Biological: hiPSC-CM therapy — 20 patients with congestive heart failure who met the inclusion and exclusion criteria will be recruited. After being fully informed and signed the informed consent, the patients will be randomly divided into two dosage groups: 100 million cells (10 patients) and 400 million cells (10 patients). Human iPSC-derived cardiomyocytes will be injected into the myocardium through a transcatheter endocardial injection system.

SUMMARY:
Heart failure is the primary cause of morbidity and mortality worldwide. Currently drug treatments for heart failure manage the symptoms, but not restore the loss cardiomyocytes due to the very limited regenerative capability in the adult heart. Novel reparative therapies that replace the cardiomyocytes loss are highly demanded to restore the cardiac function. The main purposes of this explanatory study is to investigate the safety and efficacy of the catheter-based endocardial delivery of human iPSC-derived cardiomyocytes in patients with congestive heart failure.

DETAILED DESCRIPTION:
Patients with severe congestive heart failure will be treated with allogeneic human iPSC-derived cardiomyocytes (HiCM-188) through the catheter-based injections. HiCM188, produced by Help therapeutics with cGMP condition, will be transplanted into the myocardium through a transcatheter endocardial injection system with two dosage (100 million cells or 400 million cells). The safety and efficacy assessments will be conducted at1, 3, 6 and 12 months after the cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years (including 18 and 75).
2. Signed the informed consent.
3. Patients with congestive heart failure who have received regular treatment for heart failure.
4. New York Heart Association (NYHA) Class III or IV despite optimal standard of care
5. Left Ventricular Ejection Fraction (LVEF)<40% as assessed by echocardiography ( measure in the 3 months of recruit is included, excluding the measured values within 1 month of myocardial infarction ）
6. The thickness of left ventricular ≥8mm
7. Female patient who is not pregnant or nursing during the clinical trial

Exclusion Criteria:

1. PRA ≥ 20% or DSA positive.
2. Patients received treatments such as pacemakers, ICD or CRT device.
3. Patient with severe valvular disease or presence of a mechanical valve replacement, such as PCI implantation, or patients requiring simultaneous radiofrequency ablation of atrial fibrillation.
4. Patient with any therapeutic traumatic heart surgery within 30 days.
5. Hemodynamic instability or cardiogenic shock.
6. Right heart failure.
7. Restrictive cardiomyopathy such as amyloidosis, sarcoidosis or hematochromia, constrictive pericarditis.
8. Myocardial infarction occurred within 30 days or stroke occurred within 60 days before enrollment.
9. Thickness at left ventricular free wall infarction < 6 mm.
10. Severe ventricular arrhythmias (persistent ventricular tachycardia or other conditions that the investigator considers necessary to exclude).
11. Baseline glomerular filtration rate < 30 ml/min / 1.73 m2.
12. Abnormal liver function: ALT or AST 3 times higher than the normal value.
13. Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cells count <2,500/ul or platelet count <100000 / ul.
14. Known allergies to penicillin, streptomycin or radiocontrast agent.
15. Abnormal coagulation function, INR > 1.3, which cannot be corrected.
16. Contra-indication to performance of a magnetic resonance imaging scan and PET/ECT examinations.
17. Organ transplant recipient
18. Patients with other malignant disease within 5 years prior to enrollment.
19. Non-cardiac condition that limits lifespan to < 1 year
20. On chronic therapy with immunosuppressant medication such as glucocorticoid or TNFα antagonist
21. Contra-indication to take immunosuppressant medication.
22. Serum positive for infectious diseases (HIV, HBV, HCV, TP).
23. Participated in other clinical trials within the previous 3 months .
24. Female patient who is pregnant or nursing.
25. Other condition that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major serious adverse events (SAEs) | First month post-catheterization
  Incidence of SAEs is defined as the composite of: death, fatal myocardial infarction, stroke, tamponade, cardiac perforation, ventricular arrhythmias affecting hemodynamics (> 15s), and tumorigenicity related to the hiPSC-CM .

SECONDARY OUTCOMES:
Incidence of severe arrhythmia | 1-6 months post-catheterization
  Clinically significant arrhythmias will be recorded by 24-hour ambulatory electrocardiogram
Incidence of newly formed tumors | Baseline, 1,3,6 and 12 months post-catheterization
  by comparing chest, abdominal and pelvic CT scan and PET-CT scan
Changes in penal reactive antibodies (PRA) | Baseline, 1, 3 and 6 months post-catheterization
  Changes in penal reactive antibodies (PRA) as assessed via blooddraw
Changes in donor specific antibodies (DSA) | Baseline, 1, 3 and 6 months post-catheterization
  Changes in donor specific antibodies (DSA) as assessed via blooddraw
Overall Left Ventricular systolic performance as assessed by MRI | Baseline, 1, 3, 6 and 12 months post-catheterization
  Left ventricular ejection fraction (LVEF), left ventricular end-diastolic dimension (LVEDV), left ventricular end-systolic dimension (LVESV), evaluated and compared to baseline values.
Overall Left Ventricular systolic performance as assessed by PET/ECT Scan | Baseline, 6 and 12 months post-catheterization
  Myocardial contraction and relaxation and myocardial perfusion, evaluated and compared to baseline values.
Functional status by 6 minute walk test | Baseline, 1,3,6 and 12 months post-catheterization
  valuate Functional Capacity via the Six Minute Walk Test
Functional status by New York Heart Association (NYHA) Classification | Baseline, 1,3,6 and 12 months post-catheterization
  Evaluate Functional Capacity via New York Heart Association (NYHA) Class Determination
Minnesota Living With Heart Failure Questionnaire (MLHFQ) | Baseline, 1,3,6 and 12 months post-catheterization
  Evaluate Quality Of Life Changes via Minnesota Living with Heart Failure (MLHF). The Maximum possible scores being 105 and the minimum 0. Higher scores indicate a worse or worsening quality of life, while lower scores or decreasing scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Help Therapeutics, Nanjing, Jiangsu, China